CLINICAL TRIAL: NCT07342049
Title: A Study to Determine the Safety and Performance of ConvaVAC™ Ag+ Negative Pressure Wound Therapy System in Chronic Wounds
Brief Title: ConvaVAC™ Ag+ Negative Pressure Wound Therapy System in Chronic Wounds
Acronym: ConvaVAC VLU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WC-24-452; 359501 (Other: IRAS)
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Venous Leg Ulcer (VLU)
Keywords: Venous Leg Ulcer; Negative Pressure Wound Therapy; Silver ions
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ConvaVAC Ag+ (Experimental): Negative Pressure Wound Therapy system
  Interventions: Device: ConvaVAC™ Ag+ Negative Pressure Wound Therapy System

INTERVENTIONS:
Device: ConvaVAC™ Ag+ Negative Pressure Wound Therapy System — ConvaVAC™ Ag+ Negative Pressure Wound Therapy System

SUMMARY:
Purpose of this study is to learn more about how safe and effective the ConvaVAC™ Ag+ wound therapy system is in treating certain types of long-lasting wounds, called chronic wounds. In this study, the focus is on Venous Leg Ulcers (VLUs). Chronic wounds are wounds that do not heal properly or take a long time to heal. They can cause pain, discomfort, and affect your day-to-day life. These types of wounds are also challenging for healthcare teams to treat and can take up a lot of healthcare resources. Venous Leg Ulcers (VLUs) are the most common type of chronic leg wound and affect about 1 in every 100 people. Usual treatments for VLUs include cleaning the wound, using special dressings, applying pressure (compression therapy), and sometimes using creams or dressings that contain silver to fight infection. This study is being done to see if the wound therapy system can help heal venous leg ulcers more effectively and safely.

DETAILED DESCRIPTION:
Chronic wounds, also sometimes referred to as hard-to-heal wounds, are defined as wounds that do not transition through the normal phases of healing in a timely manner. These wounds reduce health-related quality-of-life (QoL) for the patient and pose a substantial burden on healthcare professionals (HCPs) and healthcare systems. The number of chronic wounds is rising. With a global prevalence of ~1.9 per 1,000 and 1-2% in developed countries, it is predicted that the incidence of chronic wounds will increase with the aging population. Wound care accounts for 2-4% of healthcare expenditure in Europe and costs $28 billion per year in the United States.

A significant contributing factor to the delayed healing of chronic wounds is the increased risk of infection. Evidence suggests that biofilm comprises at least 78% of chronic wounds. Biofilm is communities of microorganisms embedded in a matrix of extracellular polymeric substances. This matrix protects microorganisms from antibiotics, antiseptics and the host immune response. The development of biofilm in wounds elicits a sub-optimal host inflammatory response, and is a precursor of local infection. The presence of biofilm-forming microorganisms leads to a four-fold higher chance of infection in chronic wounds compared with non-biofilm forming microorganisms (p=0.0001). The presence of biofilm in wounds can also lead to the failure of antibiotics.

Silver ions kill micro-organisms rapidly by blocking enzyme activity associated with respiration, impairing DNA synthesis and affecting cell structure. Silver is also thought to reduce bacterial adhesion and destabilize biofilm as well as increase susceptibility of bacteria to antibiotics. In recent years, a wide range of wound dressings containing elemental silver or silver releasing compounds have been developed and have gained considerable popularity. Silver dressings reduce wound healing times, hospital stays, dressing change frequency, the requirement for analgesia and reduce the number of MRSA-infected wounds. Several systematic literature reviews have been conducted highlighting the positive effects of using silver dressings on chronic wounds One of the most prevalent chronic wounds is venous leg ulcers (VLUs). Chronic leg ulcers affect around 1% (increasing to 4% in elderly populations) of the population, VLUs account for up to 90% of all chronic leg ulcers. Standard treatment of VLUs includes local wound management (e.g. debridement, moist dressings), compression therapy and topical antimicrobials. Despite standard treatment, VLUs are often associated with pain, reduced mobility, an increased risk of infection and extensive healing times. Such effects ultimately contribute to a reduced patient QoL. Only about half of VLUs heal within 4 months and recurrence rate is as high as 57% within the first year. This leaves a significant proportion of non-healing ulcers which place a burden on heath resources and patient QoL. Improvements in healing of VLUs would have a significant impact.

A promising preventative intervention is Negative Pressure Wound Therapy (NPWT), first described in the 1990's NPWT was originally designed for the treatment of open wounds. NPWT consists of a closed sealed system, the wound is covered with a foam or gauze dressing and sealed with an occlusive film. Intermittent or continuous sub-atmospheric pressure is created by a vacuum pump which draws excess fluid from the wound and collects it in a connected waste liquid collector. The system promotes granulation tissue formation, increases tissue blood flow, increases lymphatic clearance and removes bacteria from the wound bed. It therefore has the potential to improve wound outcomes rather than just manage the symptoms. NPWT has been found to be an effective treatment to heal chronic, complex and infected wounds. Recently, NPWT has been recommended in the management of chronic wounds including VLUs.

ELIGIBILITY:
Inclusion Criteria:

* A wound which is amenable to NPWT and is a VLU as defined by CEAP Classification of C6 or C6R
* Wounds that are clean or contaminated
* Wounds with at least one sign or symptom of infection
* Wounds that in the opinion of the investigator would benefit from an antimicrobial dressing
* ≥18 years old at the time of consent

Exclusion Criteria:

* Known sensitivities or allergies to components of the ConvaVAC™ Ag+ NPWT System
* Ischemic wounds with necrotic tissue or eschar present that require sharp debridement
* Wound is too small or too large based on wound dressing size (> 0.5cm2 and < 100cm2)
* Wound depth >7cm
* Wounds requiring concomitant use of DuoDERM® gel, hydrogels, petroleum-based creams/ ointment-/gels per the opinion of the investigator
* Active chemotherapy, radiation therapy, or immunotherapy for cancer or completed treatment within the last 3 months
* Any active malignancy at site of dressing application
* Exposed bone in target wound
* Exposed blood vessels or nerves in target wound
* Systemic infection and/or systemic inflammatory response syndrome (SIRS), sepsis
* Cellulitis in target wound
* Untreated deep tissue infection including but not limited to osteomyelitis, septic arthritis
* Active Pregnancy
* Subjects that in the opinion of the investigator are not suitable for enrollment
* Vulnerable subjects as determined by ICH Harmonized Guideline, Good Clinical Practice E6(R2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage area reduction (PAR) in wound size at day 14 | 14 days
  Difference between wound area at day 0 and day 14 of treatment